CLINICAL TRIAL: NCT00631202
Title: Single-Center, Open-Label, Sequential Trial to Test the Efficacy, Safety and Tolerability of Epoetin Alfa in Patients With Friedreich's Ataxia
Brief Title: Efficacy of Epoetin Alfa in Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Prof. Alessandro Filla, Dipartimento di Scienze Neurologiche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FA_EPO_3
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Friedreich's Ataxia
Keywords: FRDA; Erythropoietin; Epoetin alfa
MeSH Terms: conditions — Friedreich Ataxia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Treatment arm
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — Patients that will satisfy all inclusion/exclusion criteria will be sequentially treated with three single Epoetin alfa administrations. The first time the dose will be 600U/KG BW s.c. in a single administration. The outcome measures will be assessed. A washout period of 1 month will be necessary to eliminate any carry-over effect. A second administration of 1200U/KG BW s.c. will be performed. Outcome measures will be again assessed.
  Other Names: Eprex 40.000 IU

SUMMARY:
Friedreich's ataxia is a rare genetic disorder characterized by severe neurological disability and cardiomyopathy. Friedreich's ataxia is the consequence of frataxin deficiency. Although several drugs have been proposed, there is no available treatment. It was recently demonstrated that erythropoietin can increase the intracellular levels of frataxin in an in-vitro model.

The present project is aimed at testing the possible therapeutic approach of erythropoietin, which is an already available and commercialized drug. The investigators will perform both in-vitro and in-vivo tests, in order to asses its efficacy and safety in patients. The results will be useful to plan further clinical trials.

DETAILED DESCRIPTION:
Friedreich ataxia (FRDA) is an inherited recessive disorder characterized by progressive neurological disability. FRDA is the consequence of frataxin deficiency. Although several drugs have been proposed for FRDA, there is no available treatment. Recently it was shown that recombinant human erythropoietin (rhu-EPO) administration increases frataxin expression in cultured human lymphocytes of FRDA patients. It is therefore of primary importance to test extensively rhu-EPO's ability in increasing frataxin levels in-vitro and in-vivo. In addition rhu-EPO is an already available and commercialized drug approved for the treatment of anaemia associated with chronic renal disease, heart failure and cancer. Towards this overall purpose, we will perform an acute clinical trial in FRDA patients with rhu-EPO and will assess its effect in-vivo on frataxin expression. In addition, rhu-EPO's safety in FRDA patients based on laboratory parameters and neurological indexes will be tested. The results will be useful to gain new insight in the role of rhu-EPO in FRDA, and in the future, it may be useful to plan further clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of FA based on a homozygous GAA expansion within the FRDA with a triplet repeat sequence in the pathological range.
* Age >18, <50 years

Exclusion Criteria:

* Failure to meet one of the inclusion criteria
* Patients in treatment with Idebenone
* Wheelchair bound patients
* Significant renal, hepatic or haematological disease
* Positive history for arterial or venous thrombosis
* Acute diseases that might interfere with the study
* Positive history for arterial hypertension
* Present or programmed pregnancy
* Known hypersensitivity to study drug
* Other unacceptable concomitant medications (in particular agents thought to have a neuroprotective potential as tocopherol, amantadine, memantine, free radical scavengers).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary endpoint will be the frataxin level in PBMCs from patients at different timing from a single Epoetin alfa administration. | 0, 24, 48, 96 hours; 7, 15, 30, 60 days

SECONDARY OUTCOMES:
Echocardiography: Strain and strain rate after EPO administration at the highest study dose | 0, 30 days
Safety laboratory parameters, adverse events and tolerability | 0, 7, 15, 30, 60 days
International cooperative ataxia rating scale (ICARS). | 0, 7, 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Filla, MD, Study Director — Dipartimento di Scienze Neurologice, University "Federico II" Naples
Locations (1):
- Dipartimento di Scienze Neurologiche, Naples, Italy

REFERENCES:
- See also: Italian Ataxia association — http://www.atassia.it
- See also: University Federico II Clinics — http://www.policlinico.unina.it
- See also: University Federico II - Naples — http://www.unina.it